CLINICAL TRIAL: NCT02358941
Title: Neurofeedback and Computerized Cognitive Training in Different Settings for Children and Adolescents With Attention Deficit/Hyperactivity Disorder (ADHD)
Brief Title: Neurofeedback and Computerized Cognitive Training in Different Settings for Children and Adolescents With ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Principal Investigator, Renate Drechsler, PD Dr., University of Zurich
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SNF: 320030_149411/1
Record Dates: First submitted 2014-09-02; First posted 2015-02-09 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD, neurofeedback, computerized cognitive training, school
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Training in a school setting (Experimental): A minimum of 30 sessions (45 min.) over at least 12 weeks in the schools of the participants.
  Half of the children will be assigned to NF training, the other half to CCT.
  Interventions: Behavioral: Neurofeedback training; Behavioral: Computerized cognitive training
- Training in a clinical setting (Experimental): A minimum of 30 sessions (45 min.) over approx. 12 weeks at the Department of Child and Adolescent Psychiatry (treatment as usual).
  Half of the children will be assigned to NF training, the other half to CCT.
  Interventions: Behavioral: Neurofeedback training; Behavioral: Computerized cognitive training

INTERVENTIONS:
Behavioral: Neurofeedback training — In neurofeedback training, EEG-activity is visualized and fed back to the participant online on a computer screen. Successful regulation is rewarded by bonus points. The aim is to gain control over one's brain activity and to be able to switch to or to maintain a more wakeful, alert or focussed state.
Behavioral: Computerized cognitive training — In computerized cognitive training, impaired neuropsychological functions, such as inhibition, working memory, distractibility, are directly trained by adaptive computerized software programs. We use training programs from a scientifically based training system for patients presenting problems with sustained, focussed or selective attention, working memory, inhibition, processing speed. Good performance / improvements are rewarded with bonus points.

SUMMARY:
Attention deficit/hyperactivity disorder (ADHD) is among the most common childhood-onset psychiatric disorders, with a negative and long-lasting impact on academic achievement, social integration and quality of life. In recent years, the efficacy of non-pharmacological treatments for ADHD, such as neurofeedback training (NF) and computerized cognitive training (CCT), has been at the centre of research. Although an increasing number of well-designed studies have shown that both methods may improve ADHD core symptoms according to parents' ratings, the underlying mechanisms are still a matter of debate. Teachers often report smaller improvements, if any. This has been explained by their lesser involvement in the training. It remains questionable, however, whether other factors may also account for this effect and whether methods other than placebo control may be applied in order to demonstrate the specificity and efficacy of NF and CCT.

The main purpose of this project is to demonstrate and compare the efficacy of two different computer-based treatment methods for children and adolescents with ADHD, namely NF and CCT, and to examine the impact of different treatment settings, with half of the participants being trained in a clinical setting and the other half at school. The investigators want to show that is feasible to implement NF and CCT in a school setting and that both methods, conducted either at school or in a clinical setting, may lead to significant improvements of ADHD symptoms as well as to specific and differential effects. Besides the differential impact of the settings on informant ratings, the investigators will evaluate the effects of the training methods on neuropsychological and electrophysiological outcome. Classroom behavior of the children before and after the training will be evaluated by trained observers not informed on treatment assignments and settings.

ELIGIBILITY:
Inclusion Criteria:

* ADHD (DSM IV)

Exclusion Criteria:

* Estimated IQ < 80
* Known neurological impairment / brain injury
* Severe comorbid conditions (e.g. CD, ODD, autism)

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 102 (Actual)
Dates: Start 2013-12; Primary Completion 2017-03 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
ADHD behavioral symptoms | Outcome assessment 6 months after baseline
  Primary outcome measures will be assessed by clinical scales (Conners 3), rated by parents and teachers.

SECONDARY OUTCOMES:
Neuropsychological performance, EEG parameters | Outcome assessment 6 months after baseline
  Computerized test battery for attention and working memory; Q-EEG, event related potentials

OTHER OUTCOMES:
Classroom behavior | Observation 1 approx. 2 weeks before the start of the training, observation 2 (endpoint) approx. 2 weeks after the end of the training
  Standardized classroom observations of the participating children are conducted by a trained observer blind to whether the participant has already been trained or not and to which of the two training methods he has been allocated to.
  With regard to this measure, it is a single blind study with blinding of the assessor.

CONTACTS AND LOCATIONS:
Overall Officials: Renate Drechsler, PhD, Principal Investigator — University Clinic of Child and Adolescent Psychiatry, University of Zurich
Locations (1):
- University Clinic of Child and Adolescent Psychiatry, University of Zürich, Zurich, Switzerland

REFERENCES:
- [Derived] Minder F, Zuberer A, Brandeis D, Drechsler R. Specific Effects of Individualized Cognitive Training in Children with Attention-Deficit/Hyperactivity Disorder (ADHD): The Role of Pre-Training Cognitive Impairment and Individual Training Performance. Dev Neurorehabil. 2019 Aug;22(6):400-414. doi: 10.1080/17518423.2019.1600064. Epub 2019 Apr 25. PMID 31021250
- [Derived] Zuberer A, Minder F, Brandeis D, Drechsler R. Mixed-Effects Modeling of Neurofeedback Self-Regulation Performance: Moderators for Learning in Children with ADHD. Neural Plast. 2018 Mar 22;2018:2464310. doi: 10.1155/2018/2464310. eCollection 2018. PMID 29765401